CLINICAL TRIAL: NCT01111331
Title: Relative Bioavailability of Both BI 10773 and Warfarin and Pharmacodynamics of Warfarin After Co-administration Compared to Multiple Oral Doses of BI 10773 (25 mg Once Daily) and a Single Oral Dose of Warfarin (25 mg) Alone in Healthy Male Volunteers (an Open-label, Crossover, Clinical Phase I Study)
Brief Title: Drug Drug Interaction of Empagliflozin (BI 10773) and Warfarin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.18; 2009-018088-29 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-04-26; First posted 2010-04-27 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Warfarin

ARMS (3):
- BI 10773 25 mg (Experimental): 1 tablet 25 mg BI 10773 qd for 5 days
  Interventions: Drug: BI 10773 25 mg
- BI 10773 25 mg + Warfarin 25 mg (Experimental): 1 tablet 25 mg BI 10773 qd for 7 days plus 5 tablets 5 mg warfarin single dose
  Interventions: Drug: BI 10773 25 mg; Drug: Warfarin 25 mg
- Warfarin 25 mg (Active Comparator): 5 tablets 5 mg warfarin single dose
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: BI 10773 25 mg — 25 mg BI 10773 qd for 5 days
  Arms: BI 10773 25 mg + Warfarin 25 mg
Drug: Warfarin 25 mg — 25 mg Warfarin single dose
  Arms: BI 10773 25 mg + Warfarin 25 mg
Drug: BI 10773 25 mg — 25 mg BI 10773 qd for 12 days
  Arms: BI 10773 25 mg
Drug: Warfarin — 25 mg warfarin single dose with and without 50 mg BI 10773
  Arms: Warfarin 25 mg

SUMMARY:
The objective of the current study is to investigate the bioavailability of BI 10773 and of warfarin after concomitant multiple oral administration of BI 10773 and a single oral dose of warfarin in comparison to BI 10773 and warfarin given alone, and to investigate the pharmacodynamics of a single oral dose of warfarin with and without concomitant multiple oral administration of BI 10773.

ELIGIBILITY:
Inclusion criteria:

Healthy male subjects

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.18.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Empa / Empa Plus Warfarin / Warfarin: Patients received three treatments in the following order
  * Empagliflozin (empa) 25mg given once daily, consisting of a single tablet, on Days 1 to 5
  * Empagliflozin (empa) 25mg was given once daily on Days 1 to 7 and warfarin 25mg, consisting of 5 tablets of 5mg, was given as a single dose on Day 1
  * Warfarin 25mg was given as a single dose, consisting of 5 individual tablets, on Day 1
  There was a washout period of at least 14 days between the second and third treatment periods.
- Warfarin / Empa / Empa Plus Warfarin: Patients received three treatments in the following order
  * Warfarin 25mg was given as a single dose, consisting of 5 individual tablets, on Day 1
  * Empagliflozin (empa) 25mg given once daily, consisting of a single tablet, on Days 1 to 5
  * Empagliflozin (empa) 25mg was given once daily on Days 1 to 7 and warfarin 25mg, consisting of 5 tablets of 5mg, was given as a single dose on Day 1
  There was a washout period of at least 14 days between the first and second treatment periods.
Period: Overall Study
Arm/Group | Empa / Empa Plus Warfarin / Warfarin | Warfarin / Empa / Empa Plus Warfarin
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Overall: Total number of patients randomised and treated in the study. This was a randomised, cross-over, open-label trial consisting of three treatments. 18 patients were randomised to one of two possible treatment sequences. The three treatments were
  * Empagliflozin (empa) 25mg given once daily, consisting of a single tablet, on Days 1 to 5
  * Empagliflozin (empa) 25mg was given once daily on Days 1 to 7 and warfarin 25mg, consisting of 5 tablets of 5mg, was given as a single dose on Day 1
  * Warfarin 25mg was given as a single dose, consisting of 5 individual tablets, on Day 1
Arm/Group | Study Overall
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Empagliflozin: Area Under the Curve for the Dosing Interval at Steady State (AUCτ,ss)
Description: Area under the plasma concentration-time curve for the dosing interval τ at steady state
  In addition to the specified time frame, pre-dose samples were collected on Days 1, 3, and 4 for empa and a post-dose sample on day 1 for empa plus warfarin.
Time Frame: 0 hours (h), 20 minutes (min), 40min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h post-dose on Day 5 for for empa; 0h, 20min, 40min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 168h for empa plus warfarin.
Population: Pharmacokinetic (PK) set included all subjects who had taken at least one dose of trial medication, provided at least one observation for at least one primary PK endpoint without an important protocol violation with respect to the PK evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Empa: Empagliflozin (empa) 25mg given once daily, consisting of a single tablet, on Days 1 to 5
- Empa Plus Warfarin: Empagliflozin (empa) 25mg was given once daily on Days 1 to 7 and warfarin 25mg, consisting of 5 tablets of 5mg, was given as a single dose on Day 1
Arm/Group | Empa | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
nmol*h/L | 4580.38 (7.0) | 4621.37 (7.0)
Statistical Analysis 1: Comparison: Empa vs Empa Plus Warfarin; Ratio calculated as empa plus warfarin divided by empa; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for subject and treatment; Geometric Mean ratio = 100.89, 90% CI 2-sided [96.86 to 105.10], Standard Deviation 7.0 — Standard deviation is actually the intra-individual geometric coefficient of variation (gCV)

2. Primary Outcome: Empagliflozin: Maximum Measured Concentration at Steady State(Cmax,ss)
Description: Maximum measured plasma concentration of empagliflozin (empa) for the dosing interval τ at steady state.
  In addition to the below time frame, pre-dose samples were collected on Days 1, 3, and 4 for empa and a post-dose sample on day 1 for empa plus warfarin.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
nmol/L | 759.96 (19.9) | 764.82 (19.9)
Statistical Analysis 1: Comparison: Empa vs Empa Plus Warfarin; Ratio calculated as empa plus warfarin divided by empa; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.0021, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; Based on ANOVA with terms for subject and treatment; Geometric Mean Ratio = 100.64, 90% CI 2-sided [89.79 to 112.80], Standard Deviation 19.9 — Standard deviation is actually the intra-individual gCV

3. Primary Outcome: Warfarin R-enantiomers: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the plasma concentration-time curve from time of dosing extrapolated to infinity.
Time Frame: 0 hours (h), 20 minutes (min), 40min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 168h after administration of warfarin for both warfarin alone and warfarin plus empagliflozin
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Warfarin: Warfarin 25mg was given as a single dose, consisting of 5 individual tablets, on Day 1
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
ng*h/mL | 63585.71 (5.7) | 62626.35 (5.7)
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Ratio calculated as empa plus warfarin divided by warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 98.49, 90% CI 2-sided [95.29 to 101.80], Standard Deviation 5.7 — Standard deviation is actually the geometric coefficient of variation (gCV)

4. Primary Outcome: Warfarin R-enantiomers: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of the analyte in plasma.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
ng/mL | 1404.07 (12.4) | 1374.40 (12.4)
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Ratio calculated as empa plus warfarin divided by warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.0001, ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 97.89, 90% CI 2-sided [91.12 to 105.15], Standard Deviation 12.4 — Standard deviation is actually the geometric coefficient of variation (gCV)

5. Primary Outcome: Warfarin S-enantiomers: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the plasma concentration-time curve from time of dosing extrapolated to infinity.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
ng*h/mL | 37493.28 (4.5) | 35949.84 (4.5)
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Ratio calculated as empa plus warfarin divided by warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 95.88, 90% CI 2-sided [93.40 to 98.43], Standard Deviation 4.5 — Standard deviation is actually the intra-individual gCV

6. Primary Outcome: Warfarin S-enantiomers: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of the analyte in plasma
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
ng/mL | 1441.66 (12.7) | 1425.56 (12.7)
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Ratio calculated as empa plus warfarin divided by warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.0001, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 98.88, 90% CI 2-sided [91.84 to 106.47], Standard Deviation 12.7 — Standard deviation is actually the intra-individual gCV

7. Secondary Outcome: Empagliflozin: Plasma Concentration 24 Hours After Administration of Dose (C24,N)
Description: Plasma concentration of empagliflozin (empa) measured 24 hours after administration of the fourth dose (Cpre,5) and after the sixth dose (Cpre,7).
Time Frame: 24 hours after dose 4 or 6 respectively (day 5 and day 7)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
nmol/L
  Cpre,5 | 40.8 (33.4) | NA (NA) — Warfarin not administered
  Cpre,7 | NA (NA) — Empa alone not administered | 41.6 (36.7)

8. Secondary Outcome: Empagliflozin: Terminal Rate Constant at Steady State (λz,ss)
Description: Terminal rate constant of empagliflozin (empa) in plasma at steady state.
  In addition to the below time frame, pre-dose samples were collected on Days 1, 3, and 4 for empa and a post-dose sample on day 1 for empa plus warfarin.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Empa | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
1/h | 0.10 (10.6) | 0.10 (11.7)

9. Secondary Outcome: Empagliflozin: Terminal Half-life at Steady State (t1/2,ss)
Description: Terminal half-life of empagliflozin (empa) in plasma at steady state.
  In addition to the below time frame, pre-dose samples were collected on Days 1, 3, and 4 for empa and a post-dose sample on day 1 for empa plus warfarin.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Empa | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
h | 6.67 (10.6) | 7.07 (11.7)

10. Secondary Outcome: Empagliflozin: Time to Maximum Plasma Concentration at Steady State (Tmax,ss)
Description: Time from last dosing to maximum plasma concentration at steady state over a uniform dosing interval τ.
  In addition to the below time frame, pre-dose samples were collected on Days 1, 3, and 4 for empa and a post-dose sample on day 1 for empa plus warfarin.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Empa | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
h | 1.50 (35.0) [1.00 to 3.00] | 1.00 (55.5) [0.67 to 6.00]

11. Secondary Outcome: Empagliflozin: Mean Residence Time at Steady State After Oral Administration (MRTpo,ss)
Description: Mean residence time of empagliflozin (empa) in the body at steady state after oral administration.
  In addition to the below time frame, pre-dose samples were collected on Days 1, 3, and 4 for empa and a post-dose sample on day 1 for empa plus warfarin.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Empa | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
h | 8.64 (12.6) | 9.08 (17.5)

12. Secondary Outcome: Empagliflozin: Apparent Clearance at Steady State (CL/F,ss)
Description: Apparent clearance in plasma after extravascular administration at steady state.
  In addition to the below time frame, pre-dose samples were collected on Days 1, 3, and 4 for empa and a post-dose sample on day 1 for empa plus warfarin.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Empa | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
mL/min | 187 (14.8) | 183 (16.9)

13. Secondary Outcome: Empagliflozin: Apparent Volume of Distribution Following Extravascular Administration (Vz/F,ss)
Description: Apparent volume of distribution during the terminal phase at steady state following extravascular administration.
  In addition to the below time frame, pre-dose samples were collected on Days 1, 3, and 4 for empa and a post-dose sample on day 1 for empa plus warfarin.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Empa | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
L | 108 (8.63) | 112 (12.7)

14. Secondary Outcome: Warfarin R-enantiomers: Area Under the Curve 0 to Last Measurable Data Point (AUC0-tz)
Description: Area under the plasma concentration-time curve from time of dosing to time of last measurable data point.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
ng*h/mL | 58556.93 (5.3) | 57911.05 (5.3)
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Ratio calculated as empa plus warfarin divided by warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 98.90, 90% CI 2-sided [95.89 to 102.00], Standard Deviation 5.3 — Standard deviation is actually the geometric coefficient of variation (gCV)

15. Secondary Outcome: Warfarin R-enantiomers: Time to Maximum Plasma Concentration (Tmax)
Description: Time from dosing until maximum plasma concentration is reached
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
h | 0.84 (79.5) [0.33 to 4.00] | 1.00 (98.7) [0.33 to 7.98]

16. Secondary Outcome: Warfarin R-enantiomers: Terminal Rate Constant (λz)
Description: Terminal rate constant in plasma
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
1/h | 0.0147 (12.1) | 0.0151 (15.4)

17. Secondary Outcome: Warfarin R-enantiomers: Terminal Half-life (t1/2)
Description: Terminal half-life of the analyte in plasma
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
h | 47.1 (12.1) | 45.8 (15.4)

18. Secondary Outcome: Warfarin R-enantiomers: Mean Residence Time After Oral Administration (MRTpo)
Description: Mean residence time of the analyte in the body after oral administration
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
h | 62.9 (16.0) | 61.2 (19.1)

19. Secondary Outcome: Warfarin R-enantiomers: Apparent Clearance After Extravascular Administration (CL/F)
Description: Apparent clearance in plasma after extravascular administration
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
mL/min | 6.55 (20.8) | 6.65 (24.2)

20. Secondary Outcome: Warfarin R-enantiomers: Apparent Volume of Distribution Following Extravascular Administration (Vz/F)
Description: Apparent volume of distribution during the terminal phase λz following extravascular administration
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
L | 26.7 (15.5) | 26.4 (13.6)

21. Secondary Outcome: Warfarin S-enantiomers: Area Under the Curve 0 to Last Measurable Data Point (AUC0-tz)
Description: Area under the plasma concentration-time curve from time of dosing to time of last measurable data point.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
ng*h/mL | 36386.49 (4.4) | 34962.95 (4.4)
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Ratio calculated as empa plus warfarin divided by warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 96.09, 90% CI 2-sided [93.64 to 98.60], Standard Deviation 4.4 — Standard deviation is actually the intra-individual gCV

22. Secondary Outcome: Warfarin S-enantiomers: Time to Maximum Plasma Concentration (Tmax)
Description: Time from dosing until maximum plasma concentration is reached
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
h | 0.68 (74.6) [0.33 to 4.00] | 0.84 (85.6) [0.33 to 7.98]

23. Secondary Outcome: Warfarin S-enantiomers: Terminal Rate Constant (λz)
Description: Terminal rate constant in plasma
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
1/h | 0.0187 (13.7) | 0.0189 (12.4)

24. Secondary Outcome: Warfarin S-enantiomers: Terminal Half-life (t1/2)
Description: Terminal half-life of the analyte in plasma
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
h | 37.0 (13.7) | 36.7 (12.4)

25. Secondary Outcome: Warfarin S-enantiomers: Mean Residence Time After Oral Administration (MRTpo)
Description: Mean residence time of the analyte in the body after oral administration
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
h | 40.8 (13.8) | 38.9 (15.0)

26. Secondary Outcome: Warfarin S-enantiomers: Apparent Clearance After Extravascular Administration (CL/F)
Description: Apparent clearance in plasma after extravascular administration
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
mL/min | 11.1 (17.8) | 11.6 (16.1)

27. Secondary Outcome: Warfarin S-enantiomers: Apparent Volume of Distribution Following Extravascular Administration (Vz/F)
Description: Apparent volume of distribution during the terminal phase λz following extravascular administration
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18
L | 35.6 (21.1) | 36.8 (12.7)

28. Secondary Outcome: Warfarin: Peak International Normalised Ratio (INRmax)
Description: Peak international normalised ratio for warfarin, measured as the maximum INR over time.
Time Frame: 0 hours (h), 1h, 2h, 4h, 8h, 12h, 24h, 36h, 48h, 72h, 96h, 120h, 144h, 168h after administration of warfarin for both warfarin alone and warfarin plus empagliflozin
Population: Pharmacodynamic (PD) set included all subjects who had taken at least one dose of trial medication, provided at least one observation for at least one PD endpoint without an important protocol violation with respect to the PD evaluation.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 16 | 16
Ratio | 1.76 (NA) [1.52 to 2.05] | 1.53 (23.68) [1.32 to 1.78]
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Difference calculated as empa plus warfarin minus warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period, treatment and the baseline INR value; Geometric mean ratio = 0.87, 95% CI 2-sided [0.73 to 1.04]

29. Secondary Outcome: Warfarin: Area Under the INR-time Curve From 0 to Last Measurable Data Point (INR AUEC0-tz)
Description: Area under the concentration time curve of the INR measurements over the time interval from 0 to the time of the last quantifiable data point.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: ratio*h
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 10 | 15
ratio*h | 202.54 (NA) [185.69 to 220.91] | 178.08 (10.75) [166.63 to 190.32]
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Difference calculated as empa plus warfarin minus warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period, treatment and the baseline INR value; Geometric mean ratio = 0.88, 95% CI 2-sided [0.79 to 0.98]

30. Secondary Outcome: Warfarin: Peak International Normalised Ratio Adjusted to Baseline (INRmax,Base)
Description: Peak international normalised ratio for warfarin adjusted for baseline value (before any trial drug administration) of peak international normalised ratio
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 15 | 14
Ratio | 0.69 (NA) [0.48 to 1.01] | 0.69 (46.12) [0.46 to 1.03]
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Difference calculated as empa plus warfarin minus warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period, treatment and the baseline INR value; Geometric mean ratio = 0.99, 95% CI 2-sided [0.67 to 1.48]

31. Secondary Outcome: Warfarin: Peak Prothrombin Time (PTmax)
Description: Peak prothrombin time
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: s
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 16 | 16
s | 20.17 (NA) [18.03 to 22.56] | 18.07 (17.34) [16.15 to 20.21]
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Difference calculated as empa plus warfarin minus warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period, treatment and the baseline PT value; Geometric mean ratio = 0.90, 95% CI 2-sided [0.79 to 1.02]

32. Secondary Outcome: Warfarin: Area Under the INR-time Curve From 0 to Last Measurable Data Point Adjusted to Baseline (INR AUEC0-tz,Base)
Description: Area under the INR-time curve from time of dosing to time of last measurable data point adjusted for baseline value (before any trial drug administration) of area under the INR-time curve
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: ratio*h
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 11 | 13
ratio*h | 32.42 (NA) [18.87 to 55.69] | 36.30 (55.85) [21.44 to 61.48]
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Difference calculated as empa plus warfarin minus warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period, treatment and the baseline PT value; Geometric mean ratio = 1.12, 95% CI 2-sided [0.64 to 1.95]

33. Secondary Outcome: Warfarin: Area Under the PT-time Curve From 0 to Last Measurable Data Point (PT AUEC0-tz)
Description: Area under the PT-time curve from time of dosing to time of last measurable data point
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: s*hr
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 10 | 15
s*hr | 2508.34 (NA) [2357.25 to 2669.12] | 2281.54 (7.61) [2174.71 to 2393.62]
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Difference calculated as empa plus warfarin minus warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period, treatment and the baseline PT value; Geometric mean ratio = 0.91, 95% CI 2-sided [0.84 to 0.98]

34. Secondary Outcome: Warfarin: Peak Prothrombin Time Adjusted to Baseline (PTmax,Base)
Description: Peak prothrombin time adjusted for baseline value (before any trial drug administration) of peak prothrombin
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: s
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 15 | 14
s | 6.69 (NA) [4.74 to 9.45] | 6.51 (41.50) [4.49 to 9.42]
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Difference calculated as empa plus warfarin minus warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period, treatment and the baseline PT value; Geometric mean ratio = 0.97, 95% CI 2-sided [0.68 to 1.40]

35. Secondary Outcome: Warfarin: Area Under the PT-time Curve From 0 to Last Measurable Data Point Adjusted to Baseline (PT AUEC0-tz,Base)
Description: Area under the PT-time curve from time of dosing to time of last measurable data point adjusted for baseline value (before any trial drug administration) of area under the PT-time curve
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: s*hr
Arm/Group | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 10 | 13
s*hr | 419.24 (NA) [258.46 to 680.05] | 354.97 (54.49) [230.86 to 545.79]
Statistical Analysis 1: Comparison: Warfarin vs Empa Plus Warfarin; Difference calculated as empa plus warfarin minus warfarin; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period, treatment and the baseline PT value; Geometric mean ratio = 0.85, 95% CI 2-sided [0.47 to 1.51]

36. Secondary Outcome: Clinically Relevant Abnormalities for Physical Examination, Vital Signs, ECG, Blood Chemistry and Assessment of Tolerability by Investigator
Description: Clinically relevant abnormalities for physical examination, vital signs, ECG, blood chemistry and assessment of tolerability by investigator. New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
Time Frame: Drug administration until beginning of next sequence/end of trial, 35 days
Population: Treated set (TS) included all subjects who had taken at least one dose of trial medication.
Measure: Number; unit: participants
Arm/Group | Empa | Warfarin | Empa Plus Warfarin
Number analyzed (Participants) | 18 | 18 | 18
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Drug administration until beginning of next sequence/end of trial, 35 days
Arm/Group | Empa | Warfarin | Empa Plus Warfarin
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 4/18 | 5/18 | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa (N=18) | Warfarin (N=18) | Empa Plus Warfarin (N=18)
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Induration (General disorders) | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes